CLINICAL TRIAL: NCT07283068
Title: Intraosseous (IO) Vancomycin Into the Medial Malleolus vs Intravenous (IV) Administration in Revision Total Knee Arthroplasty (TKA)
Brief Title: IO Vancomycin Into the Medial Malleolus vs IV Administration in Revision TKA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Kwan Park, MD, Orthopedic Surgeon, The Methodist Hospital Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PRO00037463
Record Dates: First submitted 2025-12-02; First posted 2025-12-15 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Revision Total Knee Arthroplasty

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intraosseous (IO) Vancomycin (Experimental): IO vancomycin is administered via an intraosseous cannulation device (Arrow EZ-IO; Teleflex, Morrisville, NC) in the operating room after sterile preparation of the leg and draping has occurred prior to skin incision (500mg in approximately 100mL NS). Injection will take place into the medial malleolus (within a pre-specified region) immediately prior to incision.
  Interventions: Drug: Intraosseous Vancomycin
- Intravenous (IV) Vancomycin (No Intervention): Patients will receive the Houston Methodist Hospital orthopedic surgery standard of care pre-operative antibiotic regimen for revision total knee arthroplasty patients. This includes IV antibiotics (typically ancef or cefepime and vancomycin) will be started in the pre-operative period approximately 1 hour prior to incision (vancomycin dose weight based at approximately 15mg/kg [12,13] generally 1000-1750mg in 500mL NS).

INTERVENTIONS:
Drug: Intraosseous Vancomycin — IO vancomycin is administered via an intraosseous cannulation device (Arrow EZ-IO; Teleflex, Morrisville, NC) in the OR after sterile prep of the leg and draping has occurred prior to skin incision (500mg in approximately 100mL NS). Injection will take place into the medial malleolus (within a pre-specified region) immediately prior to incision.
  Arms: Intraosseous (IO) Vancomycin

SUMMARY:
Purpose of this study is to compare the efficacy of intravenous and intraosseous antibiotic administration techniques during revision total knee arthroplasty

ELIGIBILITY:
Inclusion Criteria:

* Patient is undergoing a revision total knee arthroplasty where in the opinion of the investigator, the patient's existing tibial component excludes the tibial tubercle as a valid intraosseous injection site.
* Patient is able to understand the study design and intervention and gives informed consent to participate in the study.
* Age > 18 years.

Exclusion Criteria:

* Contraindication to receiving vancomycin, cefepime, ancef, or other standard of care pre-operative antibiotic (allergy, medical issue, etc).
* Patient received or is scheduled to receive intravenous Vancomycin within 7 days prior to their planned revision procedure.
* Any hardware, condition, or anatomic status that prevents the medial malleolus from being a viable intraosseous injection site.
* Refusal to participate
* Any condition, in the opinion of the primary investigator, that deems the participant unsuitable for participation in the research study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2030-02-15 (Estimated); Study Completion 2030-06-15 (Estimated)

PRIMARY OUTCOMES:
Level of Vancomycin | During the surgery
  The study team will assess the level of vancomycin in the distal femur, proximal tibia, and systemic samples between the intravenous and intraosseous administration groups.

IPD SHARING:
Plan to Share IPD: No